CLINICAL TRIAL: NCT05403112
Title: Simultaneous Implant Placement With Autogenous Bone Ring Transplant vs Autologous Sticky Bone Graft in Maxillary Sinus Lifting " Randomization Clinical Trial"
Brief Title: Simultaneous Implant Placement With Autogenous Bone Ring
Acronym: RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Omar Saleh Ahmed Bassed (Other)
Responsible Party: Sponsor-Investigator, Omar Saleh Ahmed Bassed, Simultaneous Implant Placement With Autogenous Bone Ring Transplant vs Autologous Sticky Bone Graft in Maxillary Sinus Lifting, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Simultaneous implant placement
Record Dates: First submitted 2022-05-29; First posted 2022-06-03 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Bone Graft

STUDY DESIGN:
Intervention Model Description: randomization clinical trial
Who Masked: Care Provider
Masking Description: This trial is considered a randomized double blind clinical trial due to the following:
  1. The participant will be blinded to the technique that will be used during the surgical operation.
  2. The outcome assessor will be blinded
  3. The operator (DR.O.S.) will not be blinded for both techniques during the surgical operation, as the two techniques are different. (Dr. M.O.).
  The purpose of double blinding procedure is to reduce assessment bias and to increase accuracy and objectivity of clinical outcomes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I: autogenous bone rings (Active Comparator): sinus lifting was augmented by bone rings were harvested from chin
  Interventions: Procedure: Bone ring with open sinus lifting
- GroupII : autogenous sticky bone (Active Comparator): sinus lifting was augmented by autogenous sticky bone was harvested from chin and immediate implant placement
  Interventions: Procedure: Bone ring with open sinus lifting

INTERVENTIONS:
Procedure: Bone ring with open sinus lifting — All patients involved in this study will be divided in to two group each group will receive a different technique of sinus lifting use autogenous bone ring technique with study group and autogenous sticky bone with control group.
  Other Names: Sticky bone with open sinus lifting; simultaneous implant

SUMMARY:
This study is aiming to evaluate bone gain and secondary stability in autogenous bone ring technique using trephine bur compared to control group of sticky bone.

DETAILED DESCRIPTION:
The main prerequisite of achieving proper implant placement with ideal functional and proper restoration particularly in the posterior maxilla may compromise with violation to Schneiderian membrane especially in pneumatized maxillary Antrum when RBH < 4 mm, Conventional lateral sinus floor elevation (CLSFE) is one of the most common surgical techniques used for increasing the available bone volume to place implants and restore function and esthetics in severe atrophic maxilla.

The objective of this study was to evaluate sinus elevation with simultaneous implant placement using open technique and bone ring versus sticky bone clinically and radiographically in terms of secondary stability and bone gain around the implant

ELIGIBILITY:
Inclusion Criteria:

* Patients with edentulous vertically deficient posterior maxillary ridge a 4-5 mm. height of alveolar bone.
* Both males as well as females without any active periodontal disease.
* All patients are in a good health with no systemic, immunologic or debilitating diseases that could affect normal bone healing.
* All selected patients are non-smokers and non-alcoholics.
* Patients are free from T.M.J troubles, abnormal oral habits such as bruxism.
* The edentulous ridges are covered with optimal thickness of mucoperiosteum with no signs of inflammation, ulceration or scar tissue.
* Remaining natural teeth have good periodontal tissue support and occlusion showed sufficient inter arch space for future prosthesis.

Exclusion Criteria:

* On the local level, patients with maxillary sinus diseases, former sinus surgery and unfavorable inter maxillary relationship will be excluded.
* General contraindications to implant surgery.
* Subjected to irradiation in the head and neck area less than 1 year before implantation.
* Untreated periodontitis.
* Poor oral hygiene and motivation.
* Uncontrolled diabetes.
* Pregnant or nursing.
* Substance abuse.
* Psychiatric problems or unrealistic expectations.
* Severe bruxism or clenching.
* Immunosuppressed or immunocompromised.
* Treated or under treatment with intravenous amino-bisphosphonates.
* Lack of opposite occluding dentition/prosthesis in the area intended for implant placement.
* Active infection or severe inflammation in the area intended for implant placement.
* Need of bone augmentation procedures at implant placement.
* Unable to open mouth sufficiently to accommodate the surgical tooling.
* Patients participating in other studies, if the present protocol could not be properly followed.
* Referred only for implant placement or unable to attend a 5-year follow-up.

Ages: 26 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Change bone gain | Immediate post-operative and 6 months post-operative CT scans will be done to evaluate the bone density, apical bone gain will be measured
  bone gain (increase bone volume) Measuring the crestal bone height by CT.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Starch-Jensen T, Deluiz D, Vitenson J, Bruun NH, Tinoco EMB. Maxillary Sinus Floor Augmentation with Autogenous Bone Graft Compared with a Composite Grafting Material or Bone Substitute Alone: a Systematic Review and Meta-Analysis Assessing Volumetric Stability of the Grafting Material. J Oral Maxillofac Res. 2021 Mar 31;12(1):e1. doi: 10.5037/jomr.2021.12101. eCollection 2021 Jan-Mar. PMID 33959236
- [Result] Omara M, Abdelwahed N, Ahmed M, Hindy M. Simultaneous implant placement with ridge augmentation using an autogenous bone ring transplant. Int J Oral Maxillofac Surg. 2016 Apr;45(4):535-44. doi: 10.1016/j.ijom.2015.11.001. Epub 2015 Nov 28. PMID 26644216
- See also: Egyptian dental journal — https://edj.journals.ekb.eg/article_102929.html